CLINICAL TRIAL: NCT05000957
Title: Low Intensity Nanosecond Neodymium Laser for Complex Treatment of Pelvic Organs Prolapse
Brief Title: Pelvic Organs Prolapse Treatment Using Neodymium Laser
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: MeLSyTech, Ltd (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: POPTUNL-2021
Record Dates: First submitted 2021-07-30; First posted 2021-08-11 (Actual); Last update posted 2024-12-12 (Actual); Status verified 2024-12

CONDITIONS: Pelvic Organ Prolapse; Female Urogenital Diseases
Keywords: Pelvic Organ Prolapse; Colporrhaphy; Neodymium Laser; Laser Treatment; Nanosecond; Laser; Vaginal; Female Urogenital Diseases
MeSH Terms: conditions — Pelvic Organ Prolapse; Female Urogenital Diseases | interventions — Laser Therapy; Hematologic Tests; Electrocardiography; Vaginal Smears; Colposcopy; Ultrasonography, Doppler; Restraint, Physical

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: The treatment method cannot be hidden from the participants and the researcher because of the very different method of treatment: laser treatment followed by colporrhaphy and colporrhaphy only. However, the histologists involved in the study will not know which group the participant belongs to. The researcher will refer participants (or their materials) to these specialists, indicating their name. The Researcher will keep a document matching the participant's name and identification number.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- "Magic Max" ("Magic Gyno") Laser Treatment + Colporrhaphy (Experimental): Laser treatment of the vagina, vulva, and paraurethral region with a "Magic Max" ("Magic Gyno") laser. In total, three procedures will be performed with an interval of 4 weeks.
  During the procedure, the following sequence of actions will be performed:
  1. st Stage - vaginal processing with a conical mirror handpiece,
  2. nd Stage - vaginal processing with a corner mirror handpiece,
  3. d Stage - external vulva and paraurethral region processing with a switched beam diameter handpiece.
  A/R colporrhaphy will be performed 1 month after last laser treatment.
  Interventions: Device: Laser Treatment; Diagnostic Test: Blood analysis; Diagnostic Test: Сlinical urine test; Diagnostic Test: Electrocardiography; Diagnostic Test: Vaginal smear; Diagnostic Test: Colposcopy; Diagnostic Test: Pelvic ultrasound; Diagnostic Test: Doppler ultrasonography; Diagnostic Test: Vaginal Health Index; Diagnostic Test: Biopsy of the vaginal wall; Diagnostic Test: The Pelvic Organ Prolapse/Urinary Incontinence Sexual Questionnaire; Diagnostic Test: Pelvic Floor Distress Inventory Questionnaire; Diagnostic Test: International Consultation on Incontinence Questionnaire - Short Form; Diagnostic Test: Pelvic Floor Impact Questionnaire; Procedure: Anterior and/or posterior colporrhaphy; Other: Physical examination; Other: Сonsultation; Genetic: Buccal smear
- Colporrhaphy (control group 1) (Active Comparator): A/R colporrhaphy only will be performed.
  Interventions: Diagnostic Test: Blood analysis; Diagnostic Test: Сlinical urine test; Diagnostic Test: Electrocardiography; Diagnostic Test: Vaginal smear; Diagnostic Test: Colposcopy; Diagnostic Test: Pelvic ultrasound; Diagnostic Test: Doppler ultrasonography; Diagnostic Test: Vaginal Health Index; Diagnostic Test: Biopsy of the vaginal wall; Diagnostic Test: The Pelvic Organ Prolapse/Urinary Incontinence Sexual Questionnaire; Diagnostic Test: Pelvic Floor Distress Inventory Questionnaire; Diagnostic Test: International Consultation on Incontinence Questionnaire - Short Form; Diagnostic Test: Pelvic Floor Impact Questionnaire; Procedure: Anterior and/or posterior colporrhaphy; Other: Physical examination; Other: Сonsultation
- No Treatment (control group 2) (Other): Any surgery which do not affect condition of vagina, vulva and paraurethral region will be performed.
  Interventions: Diagnostic Test: Blood analysis; Diagnostic Test: Сlinical urine test; Diagnostic Test: Electrocardiography; Diagnostic Test: Vaginal smear; Diagnostic Test: Colposcopy; Diagnostic Test: Pelvic ultrasound; Diagnostic Test: Doppler ultrasonography; Diagnostic Test: Vaginal Health Index; Diagnostic Test: Biopsy of the vaginal wall; Diagnostic Test: The Pelvic Organ Prolapse/Urinary Incontinence Sexual Questionnaire; Diagnostic Test: Pelvic Floor Distress Inventory Questionnaire; Diagnostic Test: International Consultation on Incontinence Questionnaire - Short Form; Diagnostic Test: Pelvic Floor Impact Questionnaire; Procedure: Pelvic surgical procedure; Other: Physical examination; Other: Сonsultation

INTERVENTIONS:
Device: Laser Treatment — Laser radiation is emitted by a series of pulses following each other through a pause. The duration of one pulse is 20-200 ns, the pause between pulses is 30 us. The energy of one pulse is about 1.5 mJ.
  General laser radiation parameters for 1st and 2nd stages are: beam with diameter of 4 millimeters (mm) scans treatment area by 4 circles with step of 2 mm (50 percentage (%) overlap), average power of 10-25 Watt (W), treatment time in one point of 1-10 seconds (s), treatment step of 5 mm, from 1 to 5 repetitions of total vagina treatment. General laser radiation parameters for 3d stage are: beam diameter of 6 mm, average power of 15-30 W, duration of ns-pulses packet of 50-100 milliseconds (ms), pause between packets of 50-100 ms, treatment duration up to 65 s, treatment in permanent motion with speed of 10-50 mm/s.
  The procedure is performed without anesthesia. The doctor always focuses on the participant's feeling of warmth.
  Arms: "Magic Max" ("Magic Gyno") Laser Treatment + Colporrhaphy
Diagnostic Test: Blood analysis — Taking blood from a vein for clinical blood analysis, glucose test, hepatitis B, C viruses, human immunodeficiency viruses and syphilis test, blood clotting tests, blood type and rhesus factor determination (to include the participant in the study).
Diagnostic Test: Сlinical urine test — Urine sampling for Clinical urine test (to include the participant in the study).
Diagnostic Test: Electrocardiography — Electrocardiography investigation to determine cardiac abnormalities (to include the participant in the study).
Diagnostic Test: Vaginal smear — Vaginal smear for flora investigation, oncocytology (to include the participant in the study).
Diagnostic Test: Colposcopy — Colposcopy investigation to determine pre-malignant and malignant lesions of cervix, vagina or vulva (to include the participant in the study).
Diagnostic Test: Pelvic ultrasound — Pelvic ultrasound investigation to determine pathologies of the pelvic through a gynecological probe (to include the participant in the study).
Diagnostic Test: Doppler ultrasonography — Ultrasound investigation for assessing blood flow in the tissues of vulva region (to evaluate procedure efficiency).
Diagnostic Test: Vaginal Health Index — Vaginal Health Index will be investigated by clinical examination for vaginal elasticity, vaginal secretions, epithelial mucous membrane, vaginal hydration. Potential of hydrogen (pH) will be investigated by test-lines paper (to evaluate procedure efficiency).
Diagnostic Test: Biopsy of the vaginal wall — Sampling of the vaginal wall material in the posterior fornix area including the mucous membrane and muscle layer will be performed during colporrhaphy or any pelvic surgical procedure for histological, immunohistochemical studies, and optical coherence tomography (elastography) (to evaluate procedure efficiency)
Diagnostic Test: The Pelvic Organ Prolapse/Urinary Incontinence Sexual Questionnaire — The Pelvic Organ Prolapse/Urinary Incontinence Sexual Questionnaire will be used to collect feedback on changes in the participants' life quality (to evaluate procedure efficiency).
Diagnostic Test: Pelvic Floor Distress Inventory Questionnaire — Pelvic Floor Distress Inventory Questionnaire will be used to collect feedback on changes in the participants' life quality (to evaluate procedure efficiency).
Diagnostic Test: International Consultation on Incontinence Questionnaire - Short Form — International Consultation on Incontinence Questionnaire will be used to collect feedback on changes in the participants' life quality (to evaluate procedure efficiency).
Diagnostic Test: Pelvic Floor Impact Questionnaire — Pelvic Floor Impact Questionnaire will be used to collect feedback on changes in the participants' life quality (to evaluate procedure efficiency).
Procedure: Anterior and/or posterior colporrhaphy — Surgical procedure to repair pelvic organ prolapse followed by biopsy for histological, immunohistochemical studies, and optical coherence tomography (elastography).
  Arms: "Magic Max" ("Magic Gyno") Laser Treatment + Colporrhaphy; Colporrhaphy (control group 1)
Procedure: Pelvic surgical procedure — Any pelvic surgical procedure which do not affect condition of vagina, vulva and paraurethral region followed by biopsy for histological, immunohistochemical studies, and optical coherence tomography (elastography).
  Arms: No Treatment (control group 2)
Other: Physical examination — Pelvic examination (to include the participant in the study and observe throughout the study)
Other: Сonsultation — Сonsultation of a therapist about the absence of contraindications for surgical treatment (to include the participant in the study)
Genetic: Buccal smear — Buccal smear to performing genetic testing.
  The following markers will be analyzed:
  ESR1 rs2234693, ESR1 rs2228480, COL3A1 rs1800255, COL14A1 rs4870723, MMP9 rs3918253, MMP10 rs17435959, LOXL1 rs2304719, WNT4 rs3820282, MMP2 rs243865, TIMP2 rs2277698, CD31 / PECAM1 rs1131012, Ki67 rs11016076.
  Arms: "Magic Max" ("Magic Gyno") Laser Treatment + Colporrhaphy

SUMMARY:
The aim of this prospective study is investigation of efficiency and safety of medical device "Magic Max" ("Magic Gyno" from August 2024) for preoperative treatment of pelvic organs prolapse I-II degree of severity. To assess the condition of the vaginal walls and vulva before and after laser treatment, the following methods will be used: ultrasonography with Doppler ultrasonography, vaginal health index, histological examination, immunohistochemical examination, optical coherence tomography (OCT) (elastography). Pelvic Floor Distress Inventory Questionnaire (PFDI-20), The Pelvic Organ Prolapse/Urinary Incontinence Sexual Questionnaire (PISQ-12), International Consultation on Incontinence Questionnaire - Short Form (ICIQ-SF), Pelvic Floor Impact Questionnaire (PFIQ-7) will be used to collect feedback on changes in the participants life quality. Genetic testing of 12 gene variants will be carried out. Correlation of genes variants and treatment efficacy will be assessed. Total up to 135 participants with pelvic organs prolapse I-II degree of severity, or any other pathology of pelvic organs, which require surgical intervention will be involved in the study. Participants will be divided into three groups: group with anterior and/or posterior (A/P) colporrhaphy and laser preoperative treatment (laser treatment group), group with A/P colporrhaphy only (control group 1), and group with any other surgical intervention of pelvic area (control group 2), by 45 participants in each. The time intervals between tests will be the same for groups with A/P colporrhaphy, group with any other surgical intervention will be examined before and on the day of surgery without further observation. The main hypothesis of the study is improvement in condition of the vaginal walls after laser preoperative treatment compared with the control group 1.

DETAILED DESCRIPTION:
The principle of participant distribution into groups is the type of surgical intervention and preoperative preparation. Total up to 135 participants with pelvic organs prolapse I-II degree of severity, or any other pathology of pelvic organs, which require surgical intervention will be involved in the study. Participants will be divided into three groups: group with anterior and/or posterior (A/P) colporrhaphy and laser preoperative treatment (laser treatment group), group with A/P colporrhaphy only (control group 1), and group with any other surgical intervention of pelvic area with obtaining a biopsy of the vaginal wall (control group 2), by 45 participants in each group.

The types of examination of each group are the same and include:

General methods: physical examination, clinical blood analysis including glucose determination, clinical urine test, vaginal smear for flora and oncocytology, pelvic ultrasound, tests for hepatitis B, C viruses, human immunodeficiency viruses and syphilis, blood clotting tests, blood type and rhesus factor determination, electrocardiography, colposcopy, consultation of a therapist about the absence of contraindications for surgical treatment.

Special methods: filling out the questionnaire (Pelvic Floor Distress Inventory Questionnaire, The Pelvic Organ Prolapse/Urinary Incontinence Sexual Questionnaire, International Consultation on Incontinence Questionnaire - Short Form, Pelvic Floor Impact Questionnaire), Vaginal Health Index determination, Doppler ultrasonography of vagina, histological examination, immunohistochemical examination, optical coherence tomography (OCT) (elastography).

The treatment procedure of this study is the laser treatment of the vagina and vulva with a "Magic Max" laser ("Magic Gyno" from August 2024) with subsequent monitoring.

Genetic testing: genetic testing for the following markers will be carried out:

ESR1 rs2234693 (estrogen receptor 1), ESR1 rs2228480 (estrogen receptor 1), COL3A1 rs1800255 (collagen type III alpha 1 chain), COL14A1 rs4870723 (collagen type XIV alpha 1 chain), MMP9 rs3918253 (matrix metallopeptidase 9), MMP10 rs17435959 (matrix metallopeptidase 10), LOXL1 rs2304719 (lysyl oxidase like 1), WNT4 rs3820282 (Wnt family member 4), MMP2 rs243865 (matrix metalloproteinase type 2), TIMP2 rs2277698 (tissue inhibitor of metalloproteinase-2), CD31 / PECAM1 rs1131012 (platelet-endothelial cell adhesion molecule 1), Ki67 rs11016076 (proliferation marker Ki67).

Treatment Technique:

Laser treatment procedure will be carried out in three stages. In total, three procedures will be performed with an interval of 4 weeks. Colporrhaphy will be carried out 1 month after last treatment. Three follow-up visits will follow: 1, 6 and 12 months after colporrhaphy.

During the procedure, the following sequence of actions will be performed:

1. st Stage - vaginal processing with a conical mirror handpiece,
2. nd Stage - vaginal processing with a corner mirror handpiece,
3. rd Stage - external vulva and paraurethral region processing with a switched beam diameter handpiece.

Laser radiation is emitted by a series of pulses following each other through a pause. The duration of one pulse is 20-200 nanoseconds (ns), the pause between pulses is 30 microseconds (us). The energy of one pulse is about 1.5 millijoule (mJ). The procedure is performed without anesthesia. The doctor always focuses on the participant's feeling of warmth.

Participants of all groups will be tested with the general methods necessary to include the participant in the study at the first visit.

Control Technique:

In the control groups general surgery preparation protocol (sanitation of vagina) will be used as a therapeutic tool. After completing of preparation course, the operation will be performed.

Operation technique:

A part of the stretched vaginal wall in the posterior fornix area including the mucous membrane and muscle layer will be excised with its further suturing during colporrhaphy surgery (the excised material will be examined). This will allow comparing the vaginal walls state at the time of surgery after laser treatment and without it, and with the age norm.

Participants of all groups will be tested with the general methods necessary to include the patient in the study at the first visit.

For the laser treatment group: Studies will be carried out using filling out the questionnaires, Vaginal Health Index determination, and Doppler ultrasonography, and then laser treatment of the vagina, vulva and paraurethral region will be performed during the 2nd, 3d, and 4th visits. Filling out the questionnaires, Vaginal Health Index determination, and Doppler ultrasonography will be repeated during the 5th visit (1 month after last laser treatment and 1 day before colporrhaphy). Vaginal biopsy for histological examination, immunohistochemical examination, and optical coherence tomography (elastography) will be carried out during A/P colporrhaphy in the 6th visit. Physical examination only will be carried out during the 7th (follow-up) visit - 1 month after colporrhaphy. Filling out the questionnaires, Vaginal Health Index determination, and Doppler ultrasonography will be carried out during 8th and 9th (follow-up) visits - 6 and 12 months after colporrhaphy.

For control group 1: Studies will be carried out using filling out the questionnaires, Vaginal Health Index determination, and Doppler ultrasonography during the 1st visit after including patient. Vaginal biopsy for histological examination, immunohistochemical examination, and optical coherence tomography (elastography) will be carried out during A/P colporrhaphy in the 2nd visit. Physical examination only will be carried out during the 3th (follow-up) visit - 1 month after colporrhaphy. Filling out the questionnaire, Vaginal Health Index determination, and Doppler ultrasonography will be carried out during 4th and 5th (follow-up) visits - 6 and 12 months after colporrhaphy. Buccal smear collection will be carried out during 4th follow up visit (6 months after colporrhaphy).

Thus, a direct comparison between laser preoperational treatment and lack of preoperational treatment will be made during the investigation, 6 and 12 months after the end of each type of treatment.

For control group 2: Studies will be carried out using filling out the questionnaires, Vaginal Health Index determination, and Doppler ultrasonography during the 1st visit after including participant. Vaginal biopsy for histological examination, immunohistochemical examination, and optical coherence tomography (elastography) will be carried out during A/P colporrhaphy in the 2nd visit (no more than 1 month after 1st visit). The obtained data will allow to study the tissues of the vaginal wall in normal conditions.

The study will be carried out with the participation of several clinics:

(recruting, filling out IRC - Individual Registration Cards, buccal smear collection) (colporrhaphy and biopsy)

1. Privolzhsky Research Medical University (main scientific coordinator, histological examination, immunohistochemical examination, and optical coherence tomography (elastography)), genetic examination,
2. LLC "Medical Center" AIST "" (location of laser equipment, recruiting, filling out IRC - Individual Registration Cards laser treatment, special tests, buccal smear collection),
3. State Budgetary Institution of Health Care of the Nizhny Novgorod Region "Nizhny Novgorod Regional Clinical Oncological Dispensary" (colporrhaphy and biopsy, buccal smear collection),
4. Clinic "Preventamed", LLC "Aesthetic Medicine" (recruting, filling out IRC - Individual Registration Cards, buccal smear collection),
5. State-Funded Healthcare Institution of the Nizhny Novgorod region "Nizhny Novgorod Regional Clinical Hospital named after N.A. Semashko" (recruting, filling out IRC - Individual Registration Cards, buccal smear collection),
6. Birth house №4 of the Leninskiy District of Nizhny Novgorod named after A.F. Dobrotina (colporrhaphy and biopsy) All data obtained during the study will be transferred to the manufacturer of laser equipment "MeLSyTech" Ltd.

The study will be monitored by "MeLSyTech" Ltd as follows:

* Once a month, monitoring of provided documents (copies of individual registration records of participants, informed consent, test results) for the complete filling of the forms; the clarity of filling out forms, the possibility of systematizing information from the forms of their assessment;
* Once every six months, monitoring will be conducted with a coordinator visit of the research center and analysis activities, such as participants recruitment, data collection, data management, data analysis, reporting for adverse events, and change management;
* Once a year, the investigator submits a clinical evaluation report to the sponsor.

Statistics

The analysis will be carried out both between groups of participants receiving different types of therapy (analysis of independent groups) and within groups at different time intervals (analysis of matched groups).

Before performing statistical analysis of the data, the distribution type of the variables will be assessed. To assess the normality of distribution for each variable, histograms of frequency distributions will be visually evaluated, indicators of skewness, kurtosis, and the D'Agostino-Pearson normality test will be used.

In addition to checking the type of distribution of variables, the equality of variances of the studied groups will be assessed using the methods of analysis of variance, in particular the Brown-Forsythe test.

Methods of descriptive analysis will be used depending on the type of distribution of the variable. With a normal distribution, the mean (M) and standard deviation (SD) will be calculated. In case of an nongaussian distribution, the median (Me) and interquartile range will be calculated. Different algorithms of statistical analysis will be applied depending on the type of distribution of variables.

Comparison of the paired and unpaired groups with a normal distribution, in case of the equality of the variances, will be carried out by the methods of analysis of variance ANOVA. Comparison of groups in pairs will be performed using the post-hoc method of posterior multiple comparisons (Tukey test).

Comparison of groups in which variables do not follow the normal distribution will be carried out using the methods of nonparametric analysis of variations: the Kruskal-Wallis test (ANOVA tests) for independent groups and the Friedman test for matched groups. Dunn's multiple comparison test will be used to assess intergroup differences.

Before assessing intergroup differences, the initial samples (1 visit) will be analyzed for identity using ANOVA or nonparametric Kruskal-Wallis tests (depending on the type of data). In case of significant differences in the samples, the search and removal of extremely deviating values (outliers) will be carried out.

Differences will be considered statistically significant if the significance P values are <0.05.

ELIGIBILITY:
Inclusion Criteria:

* Age 35-50 years old;
* Participants diagnosed with pelvic organ prolapse of I-II degree of severity or any non vaginal diseases which require surgical intervention by the method of laparotomy;
* Participants were examined according to the proposed protocol;
* Participants who signed informed consent and fully informed about the purpose of the study.

Exclusion Criteria:

* Age of under 35 and over 50 years old;
* History of oncological diseases;
* Active tuberculosis;
* Inflammatory diseases of the vulva and vagina including genital herpes in the acute stage;
* Urinary tract infections;
* Damage to the vaginal mucosa;
* Pregnancy;
* Tendency to photoallergy including taking photosensitizing drugs (diuretics, antihistamines, antipsychotics);
* Porphyria;
* Cardiac deficiency of 2-3 degrees;
* Chronic renal disease;
* Diabetes mellitus (type I, II);
* Participants with greater than 2nd grade vaginal prolapse;
* Women after childbirth up to 8 weeks;
* Participants who, according to the doctor, are not able to complete the study;
* Protocol non-compliance of laser exposure sessions;
* Voluntary refusal to participate in the study;
* Violation of recommendations for the management of the period after laser treatment;
* Adverse events that occurred during laser processing and research, and associated with them.
* The occurrence of adverse events or other symptoms that are contraindications to laser procedures, as well as the occurrence of cases described in the exclusion criteria.

Ages: 35 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 129 (Actual)
Dates: Start 2021-10-03 (Actual); Primary Completion 2025-04-01 (Estimated); Study Completion 2025-04-01 (Estimated)

PRIMARY OUTCOMES:
Mean Difference from Control Groups of Collagen Fibers Thickness in Vaginal Wall | day of colporrhaphy or any surgery (laser treatment group: 1 month after last laser treatment - visit 6, control groups - no more than a month after the participant was included in the study - visit 2).
  Measurement is a part of histological examination. The quantitative assessment of collagen fibers thickness will be carried out using the ImageJ Fiji (version 1.2) software package on histological samples stained with Van Gieson's picrofuchsin. To obtain images, a light microscope with 20x objective magnification and CMOS APS-C camera will be used. The value of the collagen fiber thickness will be determined throughout the entire depth of the submucosa in 5 non-overlapping fields of view for each participant. The average value of the collagen fibers thickness will be determined based on 5 measurements in each field of view (25 measurements in total). Collagen Fibers Thickness will be measured in micrometers.
Mean Difference from Control Groups of Collagen Fibers Length in Vaginal Wall | day of colporrhaphy or any surgery (laser treatment group: 1 month after last laser treatment - visit 6, control groups - no more than a month after the participant was included in the study - visit 2).
  Measurement is a part of histological examination. The quantitative assessment of collagen fibers length will be carried out using the ImageJ Fiji (version 1.2) software package on histological samples stained with Van Gieson's picrofuchsin. To obtain images, a light microscope with 20x objective magnification and CMOS APS-C camera will be used. The value of the collagen fiber length will be determined throughout the entire depth of the submucosa in 5 non-overlapping fields of view for each participant. The average value of the collagen fiber length will be determined based on 5 measurements in each field of view (25 measurements in total). Collagen Fibers Length will be measured in micrometers.
Mean Difference from Control Groups of Thickness of the Vaginal Wall | day of colporrhaphy or any surgery (laser treatment group: 1 month after last laser treatment - visit 6, control groups - no more than a month after the participant was included in the study - visit 2).
  Measurement is a part of histological examination. Thickness of the Vaginal Wall will be measured using the ImageJ Fiji software package (version 1.2) on histological samples stained with hematoxylin and eosin. To obtain images, a light microscope with 4x objective magnification and CMOS APS-C camera will be used. The measurement will be carried out at three points of the histological section perpendicular to the surface of the epithelium. The thickness will be measured from the surface layer of the epithelium to the border of the submucosa and muscle layer. Zones of tissue deformation will not be considered. An average vaginal wall thickness will be determined for each participant. Thickness of the Vaginal Wall will be measured in millimeters (mm).

SECONDARY OUTCOMES:
Mean Change from Baseline of Artery Perfusion Index | before any intervention: laser treatment, colporrhaphy, or any surgery; before colporrhaphy - 1 month after last laser treatment (for laser treatment group); 6 and 12 months after any colporrhaphy or any surgery.
  Measurement is a part of ultrasonography. Perfusion Index will be measured with US-device. Artery Perfusion Index (API) is the total volumetric blood flow of both uterine arteries per 1 cubic centimeter (cm^3) of the uterine body. API will be calculated in percentages (%). Artery Perfusion Index is calculated by the following equation: API = (VvolRUA + VvolLUA)/Vu*100, where VvolRUA - right uterine artery volumetric blood flow (cm^3 per cardiac cycle), VvolLUA - left uterine artery volumetric blood flow (cm^3 per cardiac cycle), Vu - uterus volume (cm^3).
Mean Difference from Control Groups of Number of Fibroblasts in Vaginal Wall | day of colporrhaphy or any surgery (laser treatment group: 1 month after last laser treatment - visit 6, control groups - no more than a month after the participant was included in the study - visit 2).
  Measurement is a part of histological examination. The quantitative assessment of fibroblasts will be carried out visually in histological samples stained with hematoxylin and eosin. The number of fibroblasts will be counted for each participant in five non-overlapping fields of view at 400x magnification in view field diameter of 0.5 millimeter (mm) with light microscope. The average value will be calculated. Number of Fibroblasts will be measured in units per field of view.

OTHER OUTCOMES:
Mean Change from Baseline of Thickness of the Vaginal Wall | before any intervention: laser treatment, colporrhaphy, or any surgery; before colporrhaphy - 1 month after last laser treatment (for laser treatment group); 6 and 12 months after any colporrhaphy or any surgery.
  Measurement is a part of ultrasonography. Thickness will be measured with US-device. The vaginal probe will be inserted into the posterior fornix of the vagina, the thickness of the vaginal wall will be determined by the distance between the inner surface of the mucosa and adventitia, in millimeters (mm).
Mean Change from Baseline of Pulsatility Index of Uterine Arteries | before any intervention: laser treatment, colporrhaphy, or any surgery; before colporrhaphy - 1 month after last laser treatment (for laser treatment group); 6 and 12 months after any colporrhaphy or any surgery.
  Measurement is a part of Doppler ultrasonography. Pulsatility Index will be measured with US-device. Pulsality Index (PI) is calculated by the following equation: PI = (MSV - EDV) / (Vmean), where MSV -maximum systolic velocity, EDV - end-diastolic velocity, Vmean - mean systolic velocity. PI will be calculated in relative units.
Mean Change from Baseline of Volumetric Blood Flow of Uterine Arteries | before any intervention: laser treatment, colporrhaphy, or any surgery; before colporrhaphy - 1 month after last laser treatment (for laser treatment group); 6 and 12 months after any colporrhaphy or any surgery.
  Measurement is a part of ultrasonography. Volumetric blood flow will be measured with US-device. Volumetric blood flow (Vvol) of each uterine artery is calculated by the following equation: Vvol = Vmean * S, where Vmean - Time-averaged velocity of blood flow, S - Cross-sectional Artery Area (The S is obtained as 3.14 * (radius^2) (or its equivalent, (diameter^2)*0.785), assuming that the vessel is circular in cross-section. Volumetric blood flow will be calculated in cubic centimeters per one cardiac cycle (cc/cardiac cycle).
Mean Change from Baseline of Resistive Index of Uterine Arteries | before any intervention: laser treatment, colporrhaphy, or any surgery; before colporrhaphy - 1 month after last laser treatment (for laser treatment group); 6 and 12 months after any colporrhaphy or any surgery.
  Measurement is a part of ultrasonography. Resistive Index will be measured with US-device. The Resistive Index (RI) is calculated by the following equation: RI = (PSV - EDV) / PSV, where PSV is peak systolic velocity and EDV is end-diastolic velocity, in relative units.
Mean Change from Baseline of Vaginal Health Index Score | before any intervention: laser treatment, colporrhaphy, or any surgery; before colporrhaphy - 1 month after last laser treatment (for laser treatment group); 6 and 12 moths after any colporrhaphy or any surgery.
  Vaginal Health Index will be investigated by clinical examination for vagina:
  A. Vaginal elasticity (Characteristic=Points: Non=1, Poor=2, Fair=3, Good=4, Excellent=5), B. Vaginal secretions (None=1; Sсant, thin yellow=2; Superficial, thin white=3; Moderate, thin white=4; Normal (white)=5), C. Epithelial mucous membrane (Petechiae noted before contact=1, Bleeding with light contact=2, Bleeds with scraping, Not friable thin epithelium=4, Normal=5), D. Vaginal hydration (None, surface inflamed=1, None, surface nod inflamed=2, Minimal=3, Moderate=4, Normal=5), E. pH will be investigated by test-lines paper (≥6.1=1, 5.6-6.0=2, 5.1-5.5=3, 4.7-5.0=4, ≤4.6=5).
  Score=A+B+C+D+E
Mean Difference from Control Groups of Vascular Density in Vaginal Wall | day of colporrhaphy or any surgery (laser treatment group: 1 month after last laser treatment - visit 6, control groups - no more than a month after the participant was included in the study - visit 2).
  Measurement is a part of histological examination.The quantitative assessment of vascular density will be carried out visually on histological samples stained with hematoxylin and eosin. The number of blood vessels will be counted for each participant in five non-overlapping fields of view at 200x magnification in view field diameter of 1 mm with light microscope. The average value will be calculated. Vascular Density will be measured in units per field of view.
Mean Difference from Control Groups of Matrix Metalloproteinase-2 (MMP-2) Percentage in the Vaginal Wall | day of colporrhaphy or any surgery (laser treatment group: 1 month after last laser treatment - visit 6, control groups - no more than a month after the participant was included in the study - visit 2).
  Measurement is a part of immunohistochemical analysis. The measurement of matrix metalloproteinase-2 expression will be carried out in the vaginal wall submucosa using the ImageJ Fiji software package (version 1.2) on histological samples stained according to the instructions of the MMP-2 immunohistochemical kit. To obtain images, a light microscope with 40x objective magnification and CMOS APS-C camera will be used. Expression will be assessed semi-quantitatively in the five non-overlapping fields of view as the ratio of the positive-stained area to the field of view total area * 100. An average value will be calculated for each participant. Parameter will be measured in percentages (%).
Mean Difference from Control Groups of Tissue Inhibitor of Metalloproteinase-2 (TIMP-2) Percentage in the Vaginal Wall | day of colporrhaphy or any surgery (laser treatment group: 1 month after last laser treatment - visit 6, control groups - no more than a month after the participant was included in the study - visit 2).
  Measurement is a part of immunohistochemical analysis. The measurement of tissue inhibitor of metalloproteinase-2 expression will be carried out in the vaginal wall submucosa using the ImageJ Fiji software package (version 1.2) on histological samples stained according to the instructions of the TIMP-2 immunohistochemical kit. To obtain images, a light microscope with 40x objective magnification and CMOS APS-C camera will be used. Expression will be assessed semi-quantitatively in the five non-overlapping fields of view as the ratio of the positive-stained area to the field of view total area * 100. An average value will be calculated for each participant. Parameter will be measured in percentages (%).
Mean Difference from Control Groups of Cluster of Differentiation 31 (CD 31+) Percentage in the Vaginal Wall | day of colporrhaphy or any surgery (laser treatment group: 1 month after last laser treatment - visit 6, control groups - no more than a month after the participant was included in the study - visit 2).
  Measurement is a part of immunohistochemical analysis. The measurement of Cluster of Differentiation 31 expression will be carried out in the vaginal wall submucosa using the ImageJ Fiji software package (version 1.2) on histological samples stained according to the instructions of the CD 31+ immunohistochemical kit. To obtain images, a light microscope with 40x objective magnification and CMOS APS-C camera will be used. Expression will be assessed semi-quantitatively in the five non-overlapping fields of view as the ratio of the positive-stained area to the field of view total area * 100. An average value will be calculated for each participant. Parameter will be measured in percentages (%).
Mean Difference from Control Groups of Marker of Proliferating Cells (Ki 67) Percentage in the Vaginal Wall | day of colporrhaphy or any surgery (laser treatment group: 1 month after last laser treatment - visit 6, control groups - no more than a month after the participant was included in the study - visit 2).
  Measurement is a part of immunohistochemical analysis. The measurement of Cluster of Differentiation 31 expression will be carried out in the vaginal wall on histological samples stained according to the instructions of the Ki 67 immunohistochemical kit. Evaluation will be performed for each participant with light microscope in five non-overlapping fields of view at 400x magnification in view field diameter of 0.5 millimeter (mm). Ki 67 labeling index will be calculated for each participant as the ratio of number of positively stained cell nuclei to the total number of cell nuclei * 100. The percentage of Ki67 positive cell nuclei will be determined in regions with the most intense staining. Parameter will be measured in percentages (%).
Mean Difference from Control Groups of Stiffness of Vaginal Wall | day of colporrhaphy or any surgery (laser treatment group: 1 month after last laser treatment - visit 6, control groups - no more than a month after the participant was included in the study - visit 2).
  Elastography with optical coherence tomography (elastography) will be used to visualize inter-frame strains in the tissue and subsequently map the Young modulus. The OCT probe will slightly press onto the studied resected Vaginal Wall surface, and strain distribution in the probe vicinity will be reconstructed. For quantification of the tissue Young's modulus (stiffness), a reference silicon layer on the surface tissue with preliminary calibrated stiffness will be used. The obtained optical coherence elastography (OCE)-images are represented in the color-coded form, such that stiffer areas (those with weaker strain) are shown in blue, and soft areas, where deformation is greater, are shown in red. The Stiffness of Vaginal Wall will be measured in kiloPascal (kPa). The average stiffness value over the entire elastographic image will be obtained.
Mean Change from Baseline of "Sexual Function in Women with Urinary Incontinence and/or Pelvic Organ Prolapse" Score on Pelvic Organ Prolapse/Urinary Incontinence Sexual Questionnaire | before any intervention: laser treatment, colporrhaphy, or any surgery; before colporrhaphy - 1 month after last laser treatment (for laser treatment group); 6 and 12 months after any colporrhaphy or any surgery.
  Q1 How frequently do you feel sexual desire?Q2 Do you climax when having sexual intercourse with your partner?Q3 Do you feel sexually excited when having sexual activity with your partner?Q4 How satisfied are you with the variety of sexual activities in your sex life?Q5 Do you feel pain during sexual intercourse?Q6 Are you incontinent with sexual activity?Q7 Does fear of incontinence restrict your sexual activity?Q8 Do you avoid sexual intercourse because of bulging in the vagina?Q9 When you have sex with your partner, do you have negative emotional reactions such as fear, disgust, shame or guilt?Q10 Does your partner have a problem with erections that affects your sexual activity?Q11 Does your partner have a problem with premature ejaculation that affects your sexual activity?Q12 Compared to orgasms you have had in the past, how intense are the orgasms you have had in the past six months?Answers=Points:never(0), seldom(1), sometimes(2), usually(3), always(4).
Mean Change from Baseline of Total Score on International Consultation on Incontinence Questionnaire - Short Form | before any intervention: laser treatment, colporrhaphy, or any surgery; before colporrhaphy - 1 month after last laser treatment (for laser treatment group); 6 and 12 months after any colporrhaphy or any surgery.
  Participants answer questions:
  Q1 How often do you leak urine? Answers = Points: never (0), about once a week or less often (1), two or three times a week (2), about once a day (3), several times a day (4), all the time (5).
  Q2 How much urine do you usually leak? Answers = Points: none (0), a small amount (2), a moderate amount (4), a large amount (6)/ Q3 How much does leaking urine interfere with your everyday life? Answers = Visual Analogue Scale, where Not at all (0), A great deal (10). Total Score = Scores(Q1+Q2+Q3)
Mean Change from Baseline of "Pelvic Organ Prolapse Distress Inventory" on Pelvic Floor Distress Inventory Questionnaire | before any intervention: laser treatment, colporrhaphy, or any surgery; before colporrhaphy - 1 month after last laser treatment (for laser treatment group); 6 and 12 months after any colporrhaphy or any surgery.
  Participants answer questions:
  Q1 Do you usually experience pressure in the lower abdomen? Q2 Do you usually experience heaviness or dullness in the lower abdomen? Q3 Do you usually have a bulge or something falling out that you can see or fell in the vaginal area? Q4 Do you usually have to push on the vagina or around the rectum to have a complete bowel movement? Q5 Do you usually experience a feeling of incomplete bladder emptying? Q6 Do you ever have to push up in the vaginal area with your fingers to start or complete urination? Answers = Visual Analogue Scale, where No (0), Always bother (4). Total Score = Scores(Q1+Q2+Q3+Q4+Q5+Q6)
Mean Change from Baseline of "Colorectal-Anal Distress Inventory" on Pelvic Floor Distress Inventory Questionnaire | before any intervention: laser treatment, colporrhaphy, or any surgery; before colporrhaphy - 1 month after last laser treatment (for laser treatment group); 6 and 12 months after any colporrhaphy or any surgery.
  Participants answer questions:
  Q7 Do you feel you need to strain too hard to have a bowel movement? Q8 Do you feel you have not completely emptied your bowels at the end of a bowel movement? Q9 Do you usually lose stool beyond your control if your stool is well formed? Q10 Do you usually lose stool beyond your control if you stool is loose or liquid? Q11 Do you usually lose gas from the rectum beyond your control? Q12 Do you usually have pain when you pass your stool? Q13 Do you experience a strong sense of urgency and have to rush to the bathroom to have a bowel movement? Q14 Does part of your stool ever pass through the rectum and bulge outside during or after a bowel movement? Answers = Visual Analogue Scale, where No (0), Always bother (4). Total Score = Scores(Q7+Q8+Q9+Q10+Q11+Q12+Q13+Q14)
Mean Change from Baseline of "Urinary Distress Inventory" on Pelvic Floor Distress Inventory Questionnaire | before any intervention: laser treatment, colporrhaphy, or any surgery; before colporrhaphy - 1 month after last laser treatment (for laser treatment group); 6 and 12 months after any colporrhaphy or any surgery.
  Participants answer questions:
  Q15 Do you usually experience frequent urination Q16 Do you usually experience urine leakage associated with a feeling of urgency; that is, a strong sensation of needing to go to the bathroom? Q17 Do you usually experience urine leakage related to laughing, coughing, or sneezing? Q18 Do you usually experience small amounts of urine leakage (that is, drops)? Q19 Do you usually experience difficulty emptying your bladder? Q20 Do you usually experience pain of discomfort in the lower abdomen or genital region? Answers = Visual Analogue Scale, where No (0), Always bother (4). Total Score = Scores(Q15+Q16+Q17+Q18+Q19+Q20)
  Main Score = Total Scores("Pelvic Organ Prolapse Distress Inventory" + "Colorectal-Anal Distress Inventory" + "Urinary Distress Inventory"
Mean Change from Baseline of "Bladder or Urine" on Pelvic Floor Distress Inventory Questionnaire | before any intervention: laser treatment, colporrhaphy, or any surgery; before colporrhaphy - 1 month after last laser treatment (for laser treatment group); 6 and 12 months after any colporrhaphy or any surgery.
  Participants answer questions:
  How do symptoms or conditions of the Bladder or Urine usually affect your:
  Q1 Ability to do household chores (cooking, laundry housecleaning)? Q2 Ability to do physical activities such as walking, swimming, or other exercise? Q3 Entertainment activities such as going to a movie or concert? Q4 Ability to travel by car or bus for a distance greater than 30 minutes away from home? Q5 Participating in social activities outside your home? Q6 Emotional health (nervousness, depression, etc.)? Q7 Feeling frustrated? Answers = Not at all (0), Somewhat (1), Moderately (2), Quite a bit (3). Total Score = Mean(Q1-Q7)*100/3
Mean Change from Baseline of "Bowel or Rectum" on Pelvic Floor Distress Inventory Questionnaire | before any intervention: laser treatment, colporrhaphy, or any surgery; before colporrhaphy - 1 month after last laser treatment (for laser treatment group); 6 and 12 months after any colporrhaphy or any surgery.
  Participants answer questions:
  How do symptoms or conditions of the Bowel or Rectum usually affect your:
  Q1 Ability to do household chores (cooking, laundry housecleaning)? Q2 Ability to do physical activities such as walking, swimming, or other exercise? Q3 Entertainment activities such as going to a movie or concert? Q4 Ability to travel by car or bus for a distance greater than 30 minutes away from home? Q5 Participating in social activities outside your home? Q6 Emotional health (nervousness, depression, etc.)? Q7 Feeling frustrated? Answers = Not at all (0), Somewhat (1), Moderately (2), Quite a bit (3). Total Score = Mean(Q1-Q7)*100/3
Mean Change from Baseline of "Vagina or Pelvis" on Pelvic Floor Distress Inventory Questionnaire | before any intervention: laser treatment, colporrhaphy, or any surgery; before colporrhaphy - 1 month after last laser treatment (for laser treatment group); 6 and 12 months after any colporrhaphy or any surgery.
  Participants answer questions:
  How do symptoms or conditions of the Vagina or Pelvis usually affect your:
  Q1 Ability to do household chores (cooking, laundry housecleaning)? Q2 Ability to do physical activities such as walking, swimming, or other exercise? Q3 Entertainment activities such as going to a movie or concert? Q4 Ability to travel by car or bus for a distance greater than 30 minutes away from home? Q5 Participating in social activities outside your home? Q6 Emotional health (nervousness, depression, etc.)? Q7 Feeling frustrated? Answers = Not at all (0), Somewhat (1), Moderately (2), Quite a bit (3). Total Score = Mean(Q1-Q7)*100/3
  Main Score = Total scores("Bladder or Urine" + "Bowel or Rectum" + "Vagina or Pelvis")
Association of Marker COL3A1 rs1800255 with Changes of Collagen Fibers | 6 months after colporrhaphy.
  An analysis of marker COL3A1 rs1800255 will be carried out. An association with degree of changes collagen as a result of treatment will be assessed.
Association of Marker COL14A1 rs4870723 with Changes of Collagen Fibers | 6 months after colporrhaphy.
  An analysis of marker COL14A1 rs4870723 will be carried out. An association with degree of changes collagen as a result of treatment will be assessed.
Association of Marker ESR1 rs2234693 with Changes of Collagen Fibers | 6 months after colporrhaphy.
  An analysis of marker ESR1 rs2234693 will be carried out. An association with degree of changes collagen as a result of treatment will be assessed.
Association of Marker ESR1 rs2228480 with Changes of Collagen Fibers | 6 months after colporrhaphy.
  An analysis of marker ESR1 rs2228480 will be carried out. An association with degree of changes collagen as a result of treatment will be assessed.
Association of Marker MMP9 rs3918253 with Changes of Collagen Fibers | 6 months after colporrhaphy.
  An analysis of marker MMP9 rs3918253 will be carried out. An association with degree of changes collagen as a result of treatment will be assessed.
Association of Marker MMP10 rs17435959 with Changes of Collagen Fibers | 6 months after colporrhaphy.
  An analysis of marker MMP10 rs17435959 will be carried out. An association with degree of changes collagen as a result of treatment will be assessed.
Association of Marker LOXL1 rs2304719 with Vascular Density in Vaginal Wall | 6 months after colporrhaphy.
  An analysis of marker LOXL1 rs2304719 will be carried out. An association with degree of changes Vascular Density in Vaginal Wall as a result of treatment will be assessed.
Association of Marker LOXL1 rs2304719 with Stiffness of Vaginal Wall | 6 months after colporrhaphy.
  An analysis of marker LOXL1 rs2304719 will be carried out. An association with degree of changes Stiffness of Vaginal Wall as a result of treatment will be assessed.
Association of Marker WNT4 rs3820282 with Changes of Collagen Fibers | 6 months after colporrhaphy.
  An analysis of marker WNT4 rs3820282 will be carried out. An association with degree of changes collagen as a result of treatment will be assessed.
Association of Marker MMP2 rs243865 with Changes in Expression Level of MMP2 | 6 months after colporrhaphy.
  An analysis of marker MMP2 rs243865 will be carried out. An association with degree of changes in expression level MMP2 as a result of treatment will be assessed.
Association of Marker TIMP2 rs2277698 with Changes in Expression Level of TIMP2 | 6 months after colporrhaphy.
  An analysis of marker TIMP2 rs2277698 will be carried out. An association with degree of changes in expression level TIMP2 as a result of treatment will be assessed.
Association of Marker CD31 / PECAM1 rs1131012 with Changes in Expression Level of CD31+ | 6 months after colporrhaphy.
  An analysis of marker CD31 / PECAM1 rs 1131012 will be carried out. An association with degree of changes in expression level CD31+ as a result of treatment will be assessed.
Association of Marker Ki67 rs11016076 with Changes in Expression Level of Ki67 | 6 months after colporrhaphy.
  An analysis of marker Ki67 rs11016076 will be carried out. An association with degree of changes in expression level Ki67 as a result of treatment will be assessed.

CONTACTS AND LOCATIONS:
Overall Officials: Gennadij O Grechkanev, M.D., Principal Investigator — Privolzhsky Research Medical University
Locations (1):
- Federal State Budgetary Educational Institution of Higher Education "Privolzhsky Research Medical University" of the Ministry of Health of the Russian Federation, Nizhny Novgorod, Russia

IPD SHARING:
Plan to Share IPD: Yes
The following data can be shared with researchers upon an official request:
  The final version of the Study Protocol approved by the Local Ethics Committee; Copies of anonymized filled Individual Registration Cards (IRC); Informed Consent Form (ICF); Clinical Study Report (CSR) and/or published article (if not contradict the rules and conditions of a journal); Supplement files systematizing data.
Supporting Information: Study Protocol, ICF, CSR
Time Frame: IPD can be shared with researchers starting 3 months after CSR or article publication for five years.
Access Criteria: IPD can be shared with researchers only upon an official request from researcher's affiliation institution in the letter form on organization's letterhead paper signed by an authorized person. Official request must be directed by e-mail to the contact person (Ksenia Shatilova, shatilova@melsytech.com). The letter must contain the request purpose and statement of internal IPD use as confidential information only.
  IPD will be shared after approval by CEO of "MeLSyTech" Ltd according to the company internal rules. A requester will be notified of the decision by official letter. Depending on the decision, a requester will receive a link to the repository, or a justified rejection.